CLINICAL TRIAL: NCT01232478
Title: I Change Adherence & Raise Expectations
Acronym: iCARE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Genentech, Inc. (Industry); Cystic Fibrosis Foundation (Other); Novartis (Industry); University of Miami (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: iCARE
Record Dates: First submitted 2010-10-28; First posted 2010-11-02 (Estimated); Last update posted 2021-09-13 (Actual); Status verified 2015-03

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; Adherence; Problem-Solving; Adolescents; Education; Skills Remediation
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Comprehensive Adherence Program (CAP) (Experimental): The comprehensive adherence program emphasizes the patient's active, collaborative role in identifying adherence barriers and solving them to improve adherence to prescribed treatment regimens. Problem-solving sessions will be used to address barriers to adherence that are identified by the adolescent. The intervention also includes provision of a written, Prescribed Treatment Plan, assessment and remediation of gaps in Knowledge of Disease Management, and evaluation and re-instruction/re-training of skills needed to perform daily treatments.
  Interventions: Behavioral: Comprehensive Adherence Program (CAP)
- Standard Care (SC) (Experimental): Standard care (SC) for adolescents and young adults seen in outpatient CF clinics in Year 1 of the Study. CAP intervention during Year 2 of the Study.
  Interventions: Behavioral: Comprehensive Adherence Program (CAP)

INTERVENTIONS:
Behavioral: Comprehensive Adherence Program (CAP) — The Comprehensive Adherence Program (CAP) consists of training in the CF My Way program (a validated problem-solving adherence promotion intervention).

SUMMARY:
The iCARE study, a clustered-randomized controlled trial, is evaluating an adherence promotion intervention for adolescents that Cystic Fibrosis (CF) care teams will implement. Half the centers will receive the Comprehensive Adherence Program (CAP) for 2 years. CAP consists of training in the CF My Way program (a validated problem-solving adherence promotion intervention). The other half of the centers will receive CAP in year 2 of the study. Participants are patients age 11-20 years old who are diagnosed with CF and have been prescribed at least one of the following medications for at least 6 months prior to signing the informed consent: azithromycin, hypertonic saline, Pulmozyme®, TOBI®, or inhaled compounded tobramycin. Rate of refilling prescriptions is the primary outcome with lung function decline rates, exacerbation rates, and patient reported measures including health related quality of life and CF knowledge and skills, as secondary outcomes.

A central goal of this study is to test the effectiveness of the comprehensive adherence program (CAP), described above, versus standard care (SC) for adolescents and young adults seen in outpatient CF clinics.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients age 11 - 20 years old
* Patients with a diagnosis of CF
* Patients attend the accredited care center for regularly scheduled clinic visits
* Patient must be prescribed at least one of the following medications for at least 6 months prior to signing the informed consent:

Azithromycin Hypertonic saline Pulmozyme® TOBI® Inhaled compounded tobramycin

-Patient has consented to provide data to the CF Foundation Registry prior to conversion to PORTCFv2

Exclusion Criteria:

* Patient is planning to change care teams within the next 2 years
* Patient is seen at a satellite clinic
* Patient is on the lung transplant list (Note: participation in this study will not delay or exclude patient from being placed on the transplant list in the future or receiving a transplant once enrolled in the study)

Ages: 11 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 641 (Actual)
Dates: Start 2009-10; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Medication Adherence | 12 Months
  Medication Possession Ratio (MPR) derived from pharmacy refill records

SECONDARY OUTCOMES:
CF knowledge | 24 Months
Skills associated with CF treatments | 24 Months
Health Related Quality of Life (HRQOL) | 24 Months
  Cystic Fibrosis Questionnaire- Revised
Lung Function | 24 Months
  Forced expiratory volume in one second (FEV1) percent predicted (abstracted from CF registry)
Pulmonary exacerbation | 24 months
  IV antibiotic treatment (abstracted from CF registry)
CF hospitalizations | 24 Months
  Clinic report of pulmonary hospitalization (abstracted from CF registry)

CONTACTS AND LOCATIONS:
Overall Officials: Kristin A Riekert, PhD, Principal Investigator — Johns Hopkins University; Alexandra L Quittner, PhD, Principal Investigator — University of Miami
Locations (18):
- United States (18):
  - UAB/CHS Cystic Fibrosis Center, Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Children's Memorial Hospital, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Maine Medical Center, Portland, Maine
  - Children's Hospital Boston, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Women and Children's Hospital of Buffalo, Buffalo, New York
  - University of Rochester Medical Center, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - Akron Children's Hospital, Akron, Ohio
  - Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Toledo Children's Hospital, Toledo, Ohio
  - Primary Children's Medical Center, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
  - West Virginia University, Morgantown, West Virginia

REFERENCES:
- [Derived] Quittner AL, Eakin MN, Alpern AN, Ridge AK, McLean KA, Bilderback A, Criado KK, Chung SE, Riekert KA. Clustered randomized controlled trial of a clinic-based problem-solving intervention to improve adherence in adolescents with cystic fibrosis. J Cyst Fibros. 2019 Nov;18(6):879-885. doi: 10.1016/j.jcf.2019.05.004. Epub 2019 May 15. PMID 31103533